CLINICAL TRIAL: NCT02654509
Title: Phase 2 Open-Label Safety and Immunogenicity Study of the Eastern Equine Encephalitis (EEE) Vaccine, Inactivated, Dried, TSI-GSD 104, Lot 2-1-89, in Healthy Adult Subjects at Risk of Exposure to Eastern Equine Encephalitis Virus
Brief Title: Safety and Immunogenicity Study of the Eastern Equine Encephalitis (EEE) Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A-14568.a
Record Dates: First submitted 2016-01-11; First posted 2016-01-13 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Eastern Equine Encephalitis
MeSH Terms: conditions — Encephalomyelitis, Eastern Equine | interventions — Desiccation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EEE vaccine (Experimental): Eastern Equine Encephalitis Vaccine will be administered as primary doses of 0.5 mL given subcutaneously in the upper outer aspect of the triceps area and booster doses of 0.1 mL given intradermally in the volar aspect of the forearm. The primary series will be administered on Days 0 and 26-35 with a booster at 6 months. Titers will be collected 28-35 days after the second primary vaccine is < 1:40, the subject will receive a booster dose 28- 90 days of obtaining the titer result.
  Interventions: Biological: Eastern Equine Encephalitis Vaccine, Inactivated, Dried, TSI-GSD 104

INTERVENTIONS:
Biological: Eastern Equine Encephalitis Vaccine, Inactivated, Dried, TSI-GSD 104 — Eastern Equine Encephalitis Vaccine, Inactivated, Dried

SUMMARY:
This study is being conducted to collect safety and immunogenicity data for the Eastern Equine Encephalitis (EEE) vaccine.

DETAILED DESCRIPTION:
This study is being conducted to collect safety and immunogenicity data for the Eastern Equine Encephalitis (EEE) vaccine. To determine the frequency of adverse events in this Eastern Equine Encephalitis (EEE) vaccine study for all intent-to-treat subjects will be evaluated. Also the frequency of clinically confirmed and documented cases of Eastern Equine Encephalitis (EEE) disease among vaccinated subjects compliant with titer schedule after working with Eastern Equine Encephalitis (EEE) virus.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 to 65 years old at time of consent.
2. Have EEE virus plaque reduction neutralization 80% titers (PRNT80) < 1:20 for primary series.
3. Have EEE virus PRNT80 < 1:40 for booster series.
4. If female of childbearing potential, must agree to have a urine pregnancy test on the same day before each vaccine. (Exception: documented hysterectomy or ≥ 3 years of menopause.) The results must be negative. Females must agree not to become pregnant for 3 months after receipt of the last study treatment (vaccination).
5. Be considered at risk for exposure to EEE virus and who have submitted a Request for IND Vaccines for the EEE vaccine.
6. Sign and date the approved informed consent document and HIPAA Authorization.
7. Have in their charts:

   * medical history (including concomitant medications) within 60 days of planned first administration of vaccine
   * physical examination and laboratory tests within 1 year
   * previous chest radiograph results and electrocardiogram
8. Be medically cleared for participation by an investigator. (Examinations and/or tests may be repeated at the discretion of the principal investigator [PI].)
9. Be willing to return for all follow-up visits.
10. Agree to report any adverse events (AEs) that may or may not be associated with administration of the vaccine for at least 28 days after administration and agree to report all serious adverse events (for example, resulting in hospitalization) for the duration of the subject's participation in the study. Subjects must agree to report any pregnancy that occurs within 3 months after a vaccination.
11. Agree to defer blood, bone marrow, and organ donation for 1 year after receipt of the vaccine.

Exclusion Criteria:

1. Have completed previous EEE vaccine study as a nonresponder.
2. Have clinically significant abnormal laboratory results (including evidence of hepatitis C, hepatitis B carrier state) or elevated liver function tests (two times the normal range or at the discretion of the PI).
3. Have a personal history of an immunodeficiency or received treatment with an immunosuppressive medication, such as systemically administered glucocorticoids (eg, prednisone) within 1 month before planned administration of the vaccine or with other immunosuppressive therapies within 6 months of planned administration of the vaccine. Other immunosuppressive therapies include all cancer chemotherapeutic agents, drugs to prevent transplant rejection, interferons, monoclonal antibodies, protein kinase inhibitors, methotrexate, TNF (tumor necrosis factor) inhibitors, and any other drug determined to be immunosuppressive by the PI. Current administration of topical, inhalational, or intranasal glucocorticoids is not excluded.
4. Have confirmed HIV infection (antibody positivity).
5. Have positive pregnancy test or be a breastfeeding female.
6. Have any known allergies to components of the vaccine:

   * Neomycin sulfate
   * Formaldehyde
   * Egg
   * Human serum albumin
   * Sodium bisulfite
7. Have administration of another vaccine or investigational product within 28 days of EEE vaccination.
8. Have any unresolved AE resulting from a previous immunization.
9. Have a medical condition that, in the judgment of the PI, would impact subject safety.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2008-06-03 (Actual); Primary Completion 2016-02-16 (Actual); Study Completion 2018-03-18 (Actual)

PRIMARY OUTCOMES:
Post-Vaccination Adverse Events by System Organ Class and Severity | 30 days
  The determined adverse events after vaccination (1 month) as reported by participants by severity and system organ class.
Post-Primary Related Adverse Events by System Organ Class and Severity | 11-13 months
  The determined adverse events after primary (11-13 months) as reported by participants by severity and system organ class.
Post-Booster Related Adverse Events by System Organ Class and Severity | 1-5 weeks
  The determined adverse events after primary (1-5 weeks) as reported by participants by severity and system organ class.

SECONDARY OUTCOMES:
% vaccinated subjects with PRNT80 ≥ 1:40 after primary series. | 11-13 months
  measure immunogenicity is the 80% plaque-reduction neutralization titer (PRNT80).
% vaccinated subjects with PRNT80 ≥ 1:40 after 6-month booster dose. | 6 months
  measure immunogenicity is the 80% plaque-reduction neutralization titer (PRNT80).
% vaccinated subjects with PRNT80 ≥ 1:40 at 11-13 months after first primary dose. | 11-13 months
  measure immunogenicity is the 80% plaque-reduction neutralization titer (PRNT80).
% vaccinated subjects with PRNT80 ≥ 1:40 after week 1, 2, 3, or 4 booster doses. | 1-4 weeks
  measure immunogenicity is the 80% plaque-reduction neutralization titer (PRNT80).

OTHER OUTCOMES:
Number (%) of Vaccinated subjects with each Adverse Events. | 11-13 montms
  Adverse Event Rates by Series and Sex - Number (%) of Subjects

CONTACTS AND LOCATIONS:
Overall Officials: Robert Rivard, MD, Principal Investigator — US Army Medical Research Institute of Infectious Diseases
Locations (1):
- Special Immunizations Program, Division of Medicine, USAMRIID, Fort Deterick, Maryland, United States